CLINICAL TRIAL: NCT02250326
Title: A Phase 2, Open-Label, Multi-Center Study to Assess Safety and Efficacy of Second/Third-Line Treatment With NAB®-Paclitaxel (ABI-007) In Combination With Epigenetic Modifying Therapy Of CC-486, Or Immunotherapy of Durvalumab (MEDI4736), Or As Monotherapy In Subjects With Advanced Non-Small Cell Lung Cancer (NSCLC): Abound.2L+
Brief Title: Safety and Efficacy Study of Nab®-Paclitaxel With CC-486 or Nab®-Paclitaxel With Durvalumab, and Nab®-Paclitaxel Monotherapy as Second/Third-line Treatment for Advanced Non-small Cell Lung Cancer
Acronym: abound2L+
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-NSCL-006; 2014-001105-41 (EudraCT Number)
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Cancer of the lung; lung neoplasm; NSCLC - non-small cell lung cancer; Nonsquamou; squamous; squamous NSCLC; Tumor; locally advanced NSCLC; metastatic NSCLC; advanced lung cancer; metastatic lung cancer; non-squamous NSCLC; lung cancer; Abraxane; ABI-007; nab-paclitaxel; albumin-bound paclitaxel; taxanes; CC-486; oral azacitidine; azacitidine; second line treatment of lung cancer; second line treatment; Celgene; abound.2L; third line treatment; durvalumab; immunotherapy; MEDI4736
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms | interventions — Albumin-Bound Paclitaxel; cc-486; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Combination arm: nab-paclitaxel and CC-486 (Experimental): Subjects in the combination arm will receive nab-paclitaxel 100 mg^/m2 intravenous (IV) infusion over 30 minutes on Days 8 and 15 and CC-486 200 mg orally daily (QD) on Days 1 to14 of each 21-day treatment cycle
  Interventions: Drug: nab-paclitaxel IV; Drug: CC-486
- Monotherapy arm: nab-paclitaxel IV infusion (Experimental): Subjects in the monotherapy arm will receive nab-Paclitaxel 100 mg/m^2 IV infusion over 30 minutes on Days 1 and 8 of each 21-day treatment cycle
  Interventions: Drug: nab-paclitaxel IV
- Nab-paclitaxel and Durvalumab combination (Experimental): subjects in the nab-Paclitaxel/durvalumab combination arm will receive nab-Paclitaxel 100 mg/m2 IV infusion over 30 minutes on Days 1 and 8 and durvalumab 1125 mg IV infusion over approximately 1 hour on Day 15 of each 21-day treatment cycle
  Interventions: Drug: nab-paclitaxel IV; Drug: Duravalumab

INTERVENTIONS:
Drug: nab-paclitaxel IV — nab-Paclitaxel intravenous (IV) infusion
  Other Names: Abraxane; ABI-007
Drug: CC-486 — Oral CC-486
  Other Names: Oral AZA; Oral azacitidine
  Arms: Combination arm: nab-paclitaxel and CC-486
Drug: Duravalumab
  Arms: Nab-paclitaxel and Durvalumab combination

SUMMARY:
This is a Phase 2, open-label, multicenter study to assess the efficacy and safety of second/third-line treatment with nab-paclitaxel in combination with the epigenetic modifying therapy of CC-486 or immunotherapy of durvalumab, and nab-paclitaxel monotherapy in subjects with advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This Phase 2 study will test the hypothesis that epigenetic modifying therapy of CC-486 or immunotherapy of durvalumab can improve the anti-tumor activity of nab-paclitaxel in subjects with advanced non-small cell lung cancer (NSCLC) who have received no more than one prior chemotherapy regimen for their advanced disease. It will further assess efficacy and safety of nab-paclitaxel monotherapy in this setting. Each subject will receive study therapy as second- or third-line of treatment. Approximately 240 male and female subjects with advanced NSCLC will be assigned to one of the following treatment arms (approximately 80 subjects per group): nab-paclitaxel /CC-486 combination therapy, nab-paclitaxel/durvalumab combination therapy or nab-paclitaxel monotherapy prior to receiving first dose of Investigational Product. A permuted-block randomization method will be employed to assign the subjects among the treatment arms that are enrolling simultaneously, when applicable, stratified by the following baseline factors: ECOG performance status (0 versus 1), gender (males versus females), and smoker (yes versus no). Treatment assignments of subjects to the nab-paclitaxel/CC-486 combination therapy and nab-paclitaxel monotherapy arms will be conducted completely in a randomized fashion.

ELIGIBILITY:
Inclusion Criteria: 1.Age ≥ 18 years the time of signing the Informed Consent Form (ICF).

2. Understand and voluntarily provide written informed consent prior to the conduct of any study related assessments/procedures.

3. Able to adhere to the study visit schedule and other protocol requirements. 4. Histologically or cytologically confirmed advanced NSCLC who will receive study therapy as second- or third-line of treatment for advanced disease.

5. No other current active malignancy requiring anticancer therapy. 6. Radiographically documented measurable disease (defined by the presence of ≥ 1 radiographically documented measurable lesion).

7. One prior platinum-containing chemotherapy for metastatic or recurrent NSCLC unless patients are ineligible to receive it. Patients may have received no more than one line of chemotherapy; immunotherapy in prior line of treatment (first or second line) is allowed. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3.

8. Platelets ≥ 100,000 cells/mm3. 9. Hemoglobin (Hgb) ≥ 9 g/dL. 10. Aspartate transaminase (AST/serum glutamic oxaloacetic transaminase [SGOT]) and alanine transaminase (ALT/serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 × upper limit of normal range (ULN) or ≤ 5.0 × ULN if liver metastases.

11. Total bilirubin ≤ 1.5 ULN (unless there is a known history of Gilberts Syndrome).

12. Serum creatinine ≤ 1.5 x ULN, or calculated creatinine clearance ≥ 60 mL/min (if renal impairment is suspected 24-hour urine collection for measurement is required).

13. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1. 14. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1. 15. Females of childbearing potential [defined as a sexually mature woman who (1) have not undergone hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or (2) have not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time during the preceding 24 consecutive months)] must:

1. Have a negative pregnancy test (ß-hCG) as verified by the study doctor within 72 hours prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.
2. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting investigational product (IP), during the study therapy (including dose interruptions), and for 3 months after discontinuation of study therapy.

Male subjects must:

1. Practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 6 months following IP discontinuation, even if he has undergone a successful vasectomy.
2. Refrain from semen or sperm donation while taking durvalumab and for at least 3 months after the last dose of durvalumab.

   16. Females must abstain from breastfeeding during study participation and 3 months after IP discontinuation.

   Exclusion Criteria:
   * The presence of any of the following will exclude a subject from enrollment:

     1. Refractory to prior taxane therapy for advanced disease. Prior taxane used in the adjuvant setting does not exclude eligibility, provided there is no disease recurrence within 12 months upon completion of chemotherapy in that setting.
     2. Evidence of active brain metastases, including leptomeningeal involvement (prior evidence of brain metastasis are permitted only if asymptomatic and clinically stable for at least 8 weeks following completion of therapy). MRI of the brain (or CT scan w/contrast) is preferred.
     3. Only evidence of disease is non-measurable at study entry.
     4. Known activating EGFR mutations (such as exon 19 deletions or L858R).
     5. Known activating EML4-ALK mutations.
     6. Preexisting peripheral neuropathy of Grade > 2 (per NCI CTCAE v4.0).
     7. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
     8. Venous thromboembolism within 1 month prior to Cycle 1 Day 1.
     9. Current congestive heart failure (New York Heart Association Class II-IV).
     10. History of the following within 6 months prior to Cycle 1 Day 1: a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or clinically significant electrocardiogram (ECG) abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder.
     11. Known hepatitis B or C virus (HBV/HCV) infection, known history of human immunodeficiency virus (HIV) infection, or receiving immunosuppressive or myelosuppressive medications that would in the opinion of the investigator, increase the risk of serious neutropenic complications, history of active primary immunodeficiency, active tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice).
     12. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment.
     13. History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, or pulmonary hypersensitivity pneumonitis or multiple allergies. Any lung disease that may interfere with the detection or management of suspected drug-related pulmonary toxicity.
     14. Subject has a clinically significant malabsorption syndrome, persistent diarrhea, or known sub-acute bowel obstruction > NCI CTCAE Grade 2, despite medical management.
     15. Treatment with any chemotherapy, investigational product, biologic or hormonal therapy for cancer treatment within 28 days prior to signing the ICF. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g. hormone replacement therapy) is acceptable.
     16. History of or suspected allergy to any IP or their excipients.
     17. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
     18. Currently enrolled in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices.
     19. Any other clinically significant medical condition, psychiatric illness, and/or organ dysfunction that will interfere with the administration of the therapy according to this protocol or which, in the views of investigator, preclude combination chemotherapy.
     20. Any other malignancy within 5 years prior to randomization/treatment assignement, or advanced malignant hepatic tumors, with the exception of adequately treated squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, uteri, non-melanomatous skin cancer, carcinoma in situ of the breast, or incidental histological finding of prostate cancer (TNM Classification of Malignant Tumours (TNM) stage of T1a or T1b). (All treatment of which should have been completed 6 months prior to signing ICF).
     21. Radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting IP, and/or from whom ≥ 30% of the bone marrow was irradiated. Prior radiation therapy to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed.
     22. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
     23. Any medical condition that confounds the ability to interpret data from the study.
     24. Female patients who are pregnant or breastfeeding or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab.
     25. Male patients of reproductive potential who are not willing to employ effective birth control from screenin to 90 days after the last dose of durvalumab and from screening to 6 months after the last dose of of nab-paclitaxel.
     26. History of allogenic organ transplantation.
     27. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:
   * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection)
   * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
   * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication) 28. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of IP.

     29. Prior enrollment and treatment in a previous durvalumab clinical study. 30. Patients who have received prior anti-PD-1 or anti PD-L1:
   * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
   * All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
   * Must not have experienced a ≥ Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Subjects with endocrine AE of ≤ Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
   * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2023-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (34):
- United States (9):
  - UCSF Helen Diller Medical Center at Parnassus Heights, San Francisco, California
  - Hospital of Central Connecticut Gynecologic Oncology, New Britain, Connecticut
  - University Cancer and Blood Center, LLC, Athens, Georgia
  - Local Institution - 603, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College - New York - Presbyterian Hospital, New York, New York
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Associates in Oncology and Hematology, Chattanooga, Tennessee
  - Millennium Oncology, Houston, Texas
- Canada (2):
  - Local Institution - 642, Ottawa, Ontario
  - Local Institution - 641, Montreal, Quebec
- France (3):
  - Local Institution - 653, Lille
  - Local Institution - 651, Saint-Herblain
  - Local Institution - 652, Villejuif
- Germany (3):
  - Local Institution - 664, Essen
  - Local Institution - 663, Großhansdorf
  - Local Institution - 661, Löwenstein
- Italy (3):
  - Local Institution - 673, Bologna
  - Local Institution - 674, Parma
  - Local Institution - 672, Udine
- Spain (7):
  - Local Institution - 693, Barcelona
  - Local Institution - 695, Barcelona
  - Local Institution - 692, Madrid
  - Local Institution - 691, Madrid
  - Local Institution - 694, Málaga
  - Local Institution - 697, Valencia
  - Local Institution - 696, Valencia
- United Kingdom (7):
  - Local Institution - 630, London, Greater London
  - Local Institution - 634, Bebington, Wirral
  - Local Institution - 633, Birmingham
  - Local Institution - 635, London
  - Local Institution - 636, Manchester
  - Local Institution - 632, Newcastle upon Tyne
  - Local Institution - 631, Oxford

REFERENCES:
- [Background] Yardley DA, Coleman R, Conte P, Cortes J, Brufsky A, Shtivelband M, Young R, Bengala C, Ali H, Eakel J, Schneeweiss A, de la Cruz-Merino L, Wilks S, O'Shaughnessy J, Gluck S, Li H, Miller J, Barton D, Harbeck N; tnAcity investigators. nab-Paclitaxel plus carboplatin or gemcitabine versus gemcitabine plus carboplatin as first-line treatment of patients with triple-negative metastatic breast cancer: results from the tnAcity trial. Ann Oncol. 2018 Aug 1;29(8):1763-1770. doi: 10.1093/annonc/mdy201. PMID 29878040
- [Background] Metts JL, Alazraki AL, Clark D, Amankwah EK, Wasilewski-Masker KJ, George BA, Olson TA, Cash T. Gemcitabine/nab-paclitaxel for pediatric relapsed/refractory sarcomas. Pediatr Blood Cancer. 2018 Sep;65(9):e27246. doi: 10.1002/pbc.27246. Epub 2018 May 17. PMID 29770997
- [Background] Kim S, Signorovitch JE, Yang H, Patterson-Lomba O, Xiang CQ, Ung B, Parisi M, Marshall JL. Comparative Effectiveness of nab-Paclitaxel Plus Gemcitabine vs FOLFIRINOX in Metastatic Pancreatic Cancer: A Retrospective Nationwide Chart Review in the United States. Adv Ther. 2018 Oct;35(10):1564-1577. doi: 10.1007/s12325-018-0784-z. Epub 2018 Sep 12. PMID 30209750
- [Background] Weiss J, Gilbert J, Deal AM, Weissler M, Hilliard C, Chera B, Murphy B, Hackman T, Liao JJ, Grilley Olson J, Hayes DN. Induction chemotherapy with carboplatin, nab-paclitaxel and cetuximab for at least N2b nodal status or surgically unresectable squamous cell carcinoma of the head and neck. Oral Oncol. 2018 Sep;84:46-51. doi: 10.1016/j.oraloncology.2018.06.028. Epub 2018 Jul 19. PMID 30115475
- [Background] Cartwright TH, Parisi M, Espirito JL, Wilson TW, Pelletier C, Patel M, Babiker HM. Clinical Outcomes with First-Line Chemotherapy in a Large Retrospective Study of Patients with Metastatic Pancreatic Cancer Treated in a US Community Oncology Setting. Drugs Real World Outcomes. 2018 Sep;5(3):149-159. doi: 10.1007/s40801-018-0137-x. PMID 29946913
- [Background] Li F, Zhang H, He M, Liao J, Chen N, Li Y, Zhou S, Palmisano M, Yu A, Pai MP, Yuan H, Sun D. Different Nanoformulations Alter the Tissue Distribution of Paclitaxel, Which Aligns with Reported Distinct Efficacy and Safety Profiles. Mol Pharm. 2018 Oct 1;15(10):4505-4516. doi: 10.1021/acs.molpharmaceut.8b00527. Epub 2018 Sep 21. PMID 30180593
- [Background] Langer CJ, Kim ES, Anderson EC, Jotte RM, Modiano M, Haggstrom DE, Socoteanu MP, Smith DA, Dakhil C, Konduri K, Berry T, Ong TJ, Sanford A, Amiri K, Goldman JW, Weiss J; ABOUND.70+ Investigators. nab-Paclitaxel-Based Therapy in Underserved Patient Populations: The ABOUND.70+ Study in Elderly Patients With Advanced NSCLC. Front Oncol. 2018 Jul 24;8:262. doi: 10.3389/fonc.2018.00262. eCollection 2018. PMID 30087851
- [Background] Gajra A, Karim NA, Mulford DA, Villaruz LC, Matrana MR, Ali HY, Santos ES, Berry T, Ong TJ, Sanford A, Amiri K, Spigel DR. nab-Paclitaxel-Based Therapy in Underserved Patient Populations: The ABOUND.PS2 Study in Patients With NSCLC and a Performance Status of 2. Front Oncol. 2018 Jul 24;8:253. doi: 10.3389/fonc.2018.00253. eCollection 2018. PMID 30087850
- [Background] Pelzer U, Wislocka L, Juhling A, Striefler J, Klein F, Roemmler-Zehrer J, Sinn M, Denecke T, Bahra M, Riess H. Safety and efficacy of Nab-paclitaxel plus gemcitabine in patients with advanced pancreatic cancer suffering from cholestatic hyperbilirubinaemia-A retrospective analysis. Eur J Cancer. 2018 Sep;100:85-93. doi: 10.1016/j.ejca.2018.06.001. Epub 2018 Jul 4. PMID 30014884
- [Background] Moreno L, Casanova M, Chisholm JC, Berlanga P, Chastagner PB, Baruchel S, Amoroso L, Gallego Melcon S, Gerber NU, Bisogno G, Fagioli F, Geoerger B, Glade Bender JL, Aerts I, Bergeron C, Hingorani P, Elias I, Simcock M, Ferrara S, Le Bruchec Y, Slepetis R, Chen N, Vassal G. Phase I results of a phase I/II study of weekly nab-paclitaxel in paediatric patients with recurrent/refractory solid tumours: A collaboration with innovative therapies for children with cancer. Eur J Cancer. 2018 Sep;100:27-34. doi: 10.1016/j.ejca.2018.05.002. Epub 2018 Jun 21. PMID 29936064
- [Background] Topcul M, Ceti N IL, Ozbas Turan S, Kolusayin Ozar MO. In vitro cytotoxic effect of PARP inhibitor alone and in combination with nab-paclitaxel on triple-negative and luminal A breast cancer cells. Oncol Rep. 2018 Jul;40(1):527-535. doi: 10.3892/or.2018.6364. Epub 2018 Apr 12. PMID 29658592
- [Background] Young R, Mainwaring P, Clingan P, Parnis FX, Asghari G, Beale P, Aly A, Botteman M, Romano A, Ferrara S, Margunato-Debay S, Harris M. nab-Paclitaxel plus gemcitabine in metastatic pancreatic adenocarcinoma: Australian subset analyses of the phase III MPACT trial. Asia Pac J Clin Oncol. 2018 Oct;14(5):e325-e331. doi: 10.1111/ajco.12999. Epub 2018 Jun 22. PMID 29932294
- [Background] Neumann CCM, von Horschelmann E, Reutzel-Selke A, Seidel E, Sauer IM, Pratschke J, Bahra M, Schmuck RB. Tumor-stromal cross-talk modulating the therapeutic response in pancreatic cancer. Hepatobiliary Pancreat Dis Int. 2018 Oct;17(5):461-472. doi: 10.1016/j.hbpd.2018.09.004. Epub 2018 Sep 7. PMID 30243879
- [Background] Veenstra VL, Damhofer H, Waasdorp C, van Rijssen LB, van de Vijver MJ, Dijk F, Wilmink HW, Besselink MG, Busch OR, Chang DK, Bailey PJ, Biankin AV, Kocher HM, Medema JP, Li JS, Jiang R, Pierce DW, van Laarhoven HWM, Bijlsma MF. ADAM12 is a circulating marker for stromal activation in pancreatic cancer and predicts response to chemotherapy. Oncogenesis. 2018 Nov 16;7(11):87. doi: 10.1038/s41389-018-0096-9. PMID 30442938
- [Background] Morgensztern D, Cobo M, Ponce Aix S, Postmus PE, Lewanski CR, Bennouna J, Fischer JR, Juan-Vidal O, Stewart DJ, Fasola G, Ardizzoni A, Bhore R, Wolfsteiner M, Talbot DC, Jin Ong T, Govindan R, On Behalf Of The Abound L Investigators. ABOUND.2L+: A randomized phase 2 study of nanoparticle albumin-bound paclitaxel with or without CC-486 as second-line treatment for advanced nonsquamous non-small cell lung cancer (NSCLC). Cancer. 2018 Dec 15;124(24):4667-4675. doi: 10.1002/cncr.31779. Epub 2018 Nov 1. PMID 30383906
- [Background] Marschner N, Salat C, Soling U, Hansen R, Grebhardt S, Harde J, Nusch A, Potthoff K. Final Effectiveness and Safety Results of NABUCCO: Real-World Data From a Noninterventional, Prospective, Multicenter Study in 697 Patients With Metastatic Breast Cancer Treated With nab-Paclitaxel. Clin Breast Cancer. 2018 Dec;18(6):e1323-e1337. doi: 10.1016/j.clbc.2018.07.010. Epub 2018 Aug 10. PMID 30100104
- [Background] Watson S, de la Fouchardiere C, Kim S, Cohen R, Bachet JB, Tournigand C, Ferraz JM, Lefevre M, Colin D, Svrcek M, Meurisse A, Louvet C. Oxaliplatin, 5-Fluorouracil and Nab-paclitaxel as perioperative regimen in patients with resectable gastric adenocarcinoma: A GERCOR phase II study (FOXAGAST). Eur J Cancer. 2019 Jan;107:46-52. doi: 10.1016/j.ejca.2018.11.006. Epub 2018 Dec 7. PMID 30529902
- [Background] Li YF, Zhang C, Zhou S, He M, Zhang H, Chen N, Li F, Luan X, Pai M, Yuan H, Sun D, Li Y. Species difference in paclitaxel disposition correlated with poor pharmacological efficacy translation from mice to humans. Clin Pharmacol. 2018 Nov 8;10:165-174. doi: 10.2147/CPAA.S185449. eCollection 2018. PMID 30519122
- [Background] Hurria A, Soto-Perez-de-Celis E, Blanchard S, Burhenn P, Yeon CH, Yuan Y, Li D, Katheria V, Waisman JR, Luu TH, Somlo G, Noonan AM, Lee T, Sudan N, Chung S, Rotter A, Arsenyan A, Levi A, Choi J, Rubalcava A, Morrison R, Mortimer JE. A Phase II Trial of Older Adults With Metastatic Breast Cancer Receiving nab-Paclitaxel: Melding the Fields of Geriatrics and Oncology. Clin Breast Cancer. 2019 Apr;19(2):89-96. doi: 10.1016/j.clbc.2018.10.002. Epub 2018 Oct 16. PMID 30503309
- [Background] Fernandez A, Salgado M, Garcia A, Buxo E, Vera R, Adeva J, Jimenez-Fonseca P, Quintero G, Llorca C, Canabate M, Lopez LJ, Munoz A, Ramirez P, Gonzalez P, Lopez C, Reboredo M, Gallardo E, Sanchez-Canovas M, Gallego J, Guillen C, Ruiz-Miravet N, Navarro-Perez V, De la Camara J, Ales-Diaz I, Pazo-Cid RA, Carmona-Bayonas A. Prognostic factors for survival with nab-paclitaxel plus gemcitabine in metastatic pancreatic cancer in real-life practice: the ANICE-PaC study. BMC Cancer. 2018 Nov 29;18(1):1185. doi: 10.1186/s12885-018-5101-3. PMID 30497432
- [Background] Awasthi N, Schwarz MA, Zhang C, Schwarz RE. Augmentation of Nab-Paclitaxel Chemotherapy Response by Mechanistically Diverse Antiangiogenic Agents in Preclinical Gastric Cancer Models. Mol Cancer Ther. 2018 Nov;17(11):2353-2364. doi: 10.1158/1535-7163.MCT-18-0489. Epub 2018 Aug 30. PMID 30166402
- [Background] Cristea MC, Frankel P, Synold T, Rivkin S, Lim D, Chung V, Chao J, Wakabayashi M, Paz B, Han E, Lin P, Leong L, Hakim A, Carroll M, Prakash N, Dellinger T, Park M, Morgan RJ. A phase I trial of intraperitoneal nab-paclitaxel in the treatment of advanced malignancies primarily confined to the peritoneal cavity. Cancer Chemother Pharmacol. 2019 Mar;83(3):589-598. doi: 10.1007/s00280-019-03767-9. Epub 2019 Jan 8. PMID 30623229
- [Background] Hegewisch-Becker S, Aldaoud A, Wolf T, Krammer-Steiner B, Linde H, Scheiner-Sparna R, Hamm D, Janicke M, Marschner N; TPK-Group (Tumour Registry Pancreatic Cancer). Results from the prospective German TPK clinical cohort study: Treatment algorithms and survival of 1,174 patients with locally advanced, inoperable, or metastatic pancreatic ductal adenocarcinoma. Int J Cancer. 2019 Mar 1;144(5):981-990. doi: 10.1002/ijc.31751. Epub 2018 Oct 3. PMID 30006989
- [Background] Wang Z, Huang C, Yang JJ, Song Y, Cheng Y, Chen GY, Yan HH, Ben XS, Wang BC, Xu CR, Jiang BY, Zhou Q, Chen HJ, Wu YL. A randomised phase II clinical trial of nab-paclitaxel and carboplatin compared with gemcitabine and carboplatin as first-line therapy in advanced squamous cell lung carcinoma (C-TONG1002). Eur J Cancer. 2019 Mar;109:183-191. doi: 10.1016/j.ejca.2019.01.007. Epub 2019 Feb 7. PMID 30739019
- [Background] Barnes JA, Ellis ML, Hwang S, Emarine J, Merwin P, Salinas GD, Musher BL. Identification of Educational Gaps Among Oncologists Who Manage Patients with Pancreatic Cancer. J Gastrointest Cancer. 2019 Mar;50(1):84-90. doi: 10.1007/s12029-017-0033-8. PMID 29177608
- [Background] Woo W, Carey ET, Choi M. Spotlight on liposomal irinotecan for metastatic pancreatic cancer: patient selection and perspectives. Onco Targets Ther. 2019 Feb 21;12:1455-1463. doi: 10.2147/OTT.S167590. eCollection 2019. PMID 30863113
- [Background] Seiwert TY, Foster CC, Blair EA, Karrison TG, Agrawal N, Melotek JM, Portugal L, Brisson RJ, Dekker A, Kochanny S, Gooi Z, Lingen MW, Villaflor VM, Ginat DT, Haraf DJ, Vokes EE. OPTIMA: a phase II dose and volume de-escalation trial for human papillomavirus-positive oropharyngeal cancer. Ann Oncol. 2019 Feb 1;30(2):297-302. doi: 10.1093/annonc/mdy522. PMID 30481287
- [Background] De Luca R, Profita G, Cicero G. Nab-paclitaxel in pretreated metastatic breast cancer: evaluation of activity, safety, and quality of life. Onco Targets Ther. 2019 Feb 26;12:1621-1627. doi: 10.2147/OTT.S191519. eCollection 2019. PMID 30881017
- [Background] Morgensztern D, Ko A, O'Brien M, Ong TJ, Waqar SN, Socinski MA, Postmus PE, Bhore R. Association between depth of response and survival in patients with advanced-stage non-small cell lung cancer treated with first-line chemotherapy. Cancer. 2019 Jul 15;125(14):2394-2399. doi: 10.1002/cncr.32114. Epub 2019 Apr 1. PMID 30933354
- [Background] Li F, Yuan H, Zhang H, He M, Liao J, Chen N, Li Y, Zhou S, Palmisano M, Yu A, Pai M, Sun D. Neonatal Fc Receptor (FcRn) Enhances Tissue Distribution and Prevents Excretion of nab-Paclitaxel. Mol Pharm. 2019 Jun 3;16(6):2385-2393. doi: 10.1021/acs.molpharmaceut.8b01314. Epub 2019 May 1. PMID 31002261
- [Background] Sonbol MB, Ahn DH, Goldstein D, Okusaka T, Tabernero J, Macarulla T, Reni M, Li CP, O'Neil B, Van Cutsem E, Bekaii-Saab T. CanStem111P trial: a Phase III study of napabucasin plus nab-paclitaxel with gemcitabine. Future Oncol. 2019 Apr;15(12):1295-1302. doi: 10.2217/fon-2018-0903. Epub 2019 Feb 15. PMID 30768369
- [Derived] Morgensztern D, Dols MC, Ponce Aix S, Postmus PE, Bennouna J, Fischer JR, Juan-Vidal O, Stewart DJ, Ardizzoni A, Bhore R, Wolfsteiner M, Reck M, Talbot D, Govindan R, Ong TJ. nab-Paclitaxel Plus Durvalumab in Patients With Previously Treated Advanced Stage Non-small Cell Lung Cancer (ABOUND.2L+). Front Oncol. 2021 Feb 11;10:569715. doi: 10.3389/fonc.2020.569715. eCollection 2020. PMID 33643895
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants included those with advanced non-small cell lung cancer who had received no more than one prior containing chemotherapy regimen. Immunotherapy as a prior line of treatment was allowed. Randomization was stratified by eastern cooperative oncology group performance status, gender and the smoking status of the participant.
Groups:
- Nab-Paclitaxel + CC-486: Participants received nab-paclitaxel 100 mg/m^2 by intravenous (IV) infusion over 30 minutes on Days 8 and 15. CC-486 200 mg tablets on Days 1 to 14 of each 21-day treatment cycle until disease progression (DP), development of an unacceptable toxicity, death, lost to follow-up, or withdrawal of consent, in accordance with local standard of care.
- Nab-Paclitaxel + Durvalumab: Participants received nab-paclitaxel 100 mg/m^2 by IV infusion over 30 minutes on Days 1 and 8. Durvalumab (durva) 1125 mg/m^2 by IV infusion over 1 hour on Day 15 of each 21-day treatment cycle until disease progression, development of an unacceptable toxicity, death, lost to follow-up, or withdrawal of consent, in accordance with local standard of care.
- Nab-Paclitaxel: Participants received nab-paclitaxel 100 mg/m^2 by IV infusion over 30 minutes on Days 1 and 8 each 21-day treatment cycle until disease progression, development of an unacceptable toxicity, death, lost to follow-up, or withdrawal of consent, in accordance with local standard of care.
Period: Pre-treatment
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel
Started (Started = Randomized) | 81 | 79 | 80
Completed (Completed = Treated) | 79 | 78 | 79
Not Completed | 2 | 1 | 1
Period: Treatment
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel
Started | 79 | 78 | 79
Completed | 0 | 0 | 0
Not Completed | 79 | 78 | 79
Not completed — Death | 1 | 13 | 2
Not completed — Adverse Event | 8 | 8 | 9
Not completed — Progressive Disease | 42 | 40 | 47
Not completed — Symptomatic Deterioration | 9 | 4 | 10
Not completed — Withdrawal by Subject | 11 | 6 | 4
Not completed — Other reasons | 8 | 7 | 7
Period: Extension Period
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel
Started (Started = met the criteria for treatment continuation in the extension period) | 0 | 4 (Participants who continued to benefit from study treatment with nab-paclitaxel and/or durvalumab, without unacceptable toxicities) | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 4 | 0
Not completed — Progressive Disease | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Withdrawal by investigator | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population included all assigned participants regardless of whether the participant received any investigational product (IP) or had any efficacy assessments performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel | Total
Number analyzed (Participants) | 81 | 79 | 80 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.00) | 62.7 (10.74) | 62.6 (9.58) | 63.1 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 30 | 86
  Male | 50 | 54 | 50 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 3 | 10
  Not Hispanic or Latino | 67 | 73 | 66 | 206
  Unknown or Not Reported | 13 | 0 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 67 | 77 | 63 | 207
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 14 | 1 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Kaplan Meier Estimate of Progression-Free Survival (PFS) as Assessed by the Investigator
Description: Progression-free survival was defined as the time in months from the date of randomization/assignment to the date of disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria documented by computed tomography (CT) scan, not including symptomatic deterioration, or death (any cause) on or prior to the clinical cut-off date, which ever occurred earlier. Participants who did not have disease progression and had not died, regardless of whether they were discontinued from treatment, were censored at the date of last tumor assessment, on or prior to the clinical cut-off date that the participant was progression free. Progressive Disease was defined as at least a 20% increase in the sum of diameters of target lesions from nadir.
Time Frame: From date of first dose of IP to DP; up to data cut-off date of 30 August (Aug) 2017 for nab-paclitaxel and CC-486 + nab-paclitaxel and 23 December (Dec) 2017 for Durva + nab-paclitaxel; participants were followed for PFS for up to 18 months
Population: Intent to Treat Population included all randomized or assigned participants regardless of whether the participant received any study drug or had any efficacy assessments performed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Nab-Paclitaxel Alone: Participants received nab-paclitaxel 100 mg/m^2 by intravenous infusion over 30 minutes on Days 1 and 8 each 21-day treatment cycle until disease progression, development of an unacceptable toxicity, death, lost to follow-up, or withdrawal of consent, in accordance with local standard of care.
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel Alone
Number analyzed (Participants) | 81 | 79 | 80
months | 3.2 [2.30 to 4.30] | 4.5 [3.45 to 5.88] | 4.2 [2.79 to 5.06]
Statistical Analysis 1: Comparison: Nab-Paclitaxel + CC-486 vs Nab-Paclitaxel Alone; Based on stratified Cox proportional hazards regression model; Test type: Superiority; Based on stratification factors of ECOG Performance Status (0 or 1), sex (male or female), and current smoker status (yes or no); Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.90 to 1.94]

2. Secondary Outcome: Percentage of Participants Who Achieved a Complete Response (CR), Partial Response (PR) or Stable Disease (SD) According to RECIST V 1.1 Criteria
Description: Disease control rate was defined as the percentage of participants who had a CR, PR or SD during the course of the study, according to RECIST version 1.1 criteria, as evaluated by the investigator. RECIST Version 1.1 criteria is defined as follows: - Complete Response is the disappearance of all target lesions; - Partial Response is at least a 30% decrease in the sum of diameters of target lesions from baseline; - Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for progressive disease. Responses were evaluated every 6 weeks.
Time Frame: Up to 30 Aug 2017 for nab-paclitaxel and CC-486 + nab-paclitaxel and 23 Dec 2017 for Durva + nab-paclitaxel; maximum treatment duration = 82.1 weeks, 52.6 weeks and 66.1 weeks for nab-paclitaxel, CC-486 + nab-paclitaxel and Durva + nab-paclitaxel
Population: ITT Population included all randomized or assigned participants regardless of whether the participant received any study drug or had any efficacy assessments performed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel Alone
Number analyzed (Participants) | 81 | 79 | 80
Percentage of Participants | 65.4 [54.0 to 75.7] | 70.9 [59.6 to 80.6] | 67.5 [56.1 to 77.6]
Statistical Analysis 1: Comparison: Nab-Paclitaxel + CC-486 vs Nab-Paclitaxel Alone; Test type: Superiority; Disease Control Rate Ratio = 0.97, 95% CI 2-sided [0.778 to 1.207] — 95% CI was calculated using Clopper-Pearson method; Direction of Disease Control Rate Ratio is DCR of Nab-Paclitaxel + CC-486 Combination Arm over DCR of Nab-Paclitaxel Alone

3. Secondary Outcome: Percentage of Participants Who Achieved a Best Overall Response of Complete Response or Partial Response According to RECIST V 1.1 Criteria
Description: Overall Response was defined as percentage of participants who achieved a radiologic confirmed complete response or partial response according to RECIST V 1.1 criteria and compared with baseline among all tumor assessments, where baseline was the last CT obtained prior to or on Day 1 of treatment. Per RECIST V 1.1 criteria, a CR is defined as a disappearance of all target lesions; a PR is defined as having at least a 30% decrease in the sum of diameters of target lesions from baseline. Responses were evaluated every 6 weeks.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel Alone
Number analyzed (Participants) | 81 | 79 | 80
percentage of participants | 13.6 [7.0 to 23.0] | 27.8 [18.3 to 39.1] | 16.3 [8.9 to 26.2]
Statistical Analysis 1: Comparison: Nab-Paclitaxel + CC-486 vs Nab-Paclitaxel Alone; Test type: Superiority; Overall Response Rate Ratio = 0.84, 95% CI 2-sided [0.398 to 1.754] — 95% CI was calculated using Clopper-Pearson method; Direction of Overall Response Rate Ratio is ORR of Nab-Paclitaxel + CC-486 Combination Arm over ORR of nab-Paclitaxel Alone

4. Secondary Outcome: Kaplan Meier Estimate of Overall Survival (OS)
Description: Overall survival was defined as the time in months between randomization/treatment assignment and death from any cause. Participants who were still alive as of the clinical cut-off date had their OS censored at the date of last contact or clinical cut-off, whichever was earlier. Participants who were lost to follow-up prior to the end of the study or who were withdrawn from the study were censored at the time of last contact.
Time Frame: Up to 30 Aug 2017 for nab-paclitaxel and CC-486 + nab-paclitaxel and 23 Dec 2017 for Durva + nab-paclitaxel; participants were followed for overall survival up to 30 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel Alone
Number analyzed (Participants) | 81 | 79 | 80
Months | 8.1 [6.64 to 11.86] | 10.1 [7.75 to NA] — The 95% CI upper bound of the median OS time is not estimable, because the survival rate is greater than 40% for all values of time, therefore, no time that corresponding to the 40% survival rate and below. | 17.0 [8.21 to NA] — The 95% CI upper bound of the median OS time is not estimable, because the survival rate is greater than 40% for all values of time, therefore, no time that corresponding to the 40% survival rate and below.
Statistical Analysis 1: Comparison: Nab-Paclitaxel + CC-486 vs Nab-Paclitaxel Alone; Based on stratified Cox proportional hazards regression model; Test type: Superiority; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.7, 95% CI 2-sided [1.08 to 2.57]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) During the Entire Treatment Period
Description: TEAEs were defined as any adverse event or serious adverse event that occurred or worsened on or after the day of the first dose of the IP through 28 days after the last dose of IP for Arms A and C or up to 90 days after the last dose for Arm B, and those SAEs made known to the investigator at any time thereafter that are suspected of being related to IP. A serious AE (SAE) = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs were graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 and the scale: Grade 1 = Mild l intervention/therapy required Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Death.
Time Frame: TEAEs were collected up to 4 weeks after receiving last dose of investigational product (IP) for nab-paclitaxel and CC-486 + nab-paclitaxel, and up to 90 days after the last IP dose for Durva + nab-paclitaxel; TEAEs were collected up to 354 weeks
Population: Safety Population included all participants who were randomized and received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Nab-Paclitaxel: Participants received nab-paclitaxel 100 mg/m^2 by intravenous infusion over 30 minutes on Days 1 and 8 each 21-day treatment cycle until disease progression, development of an unacceptable toxicity, death, lost to follow-up, or withdrawal of consent, in accordance with local standard of care.
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel
Number analyzed (Participants) | 79 | 78 | 79
Participants
  TEAE | 79 | 78 | 78
  Serious TEAE | 30 | 44 | 30
  Grade (GR) 3/4 TEAE | 48 | 57 | 47
  Grade 3 or Higher | 49 | 59 | 47
  Treatment Related TEAE | 74 | 72 | 68
  Treatment Related Serious TEAE | 11 | 20 | 5
  Treatment Related GR 3 or Higher TEAE | 32 | 36 | 25
  TEAE With Action to Reduce/Interrupt IP | 49 | 59 | 38
  Treatment-Related to Reduce or Interrupt IP | 36 | 36 | 27
  TEAE with Action Taken to Withdraw IP | 8 | 11 | 9
  Treatment Related TEAE with Action Taken to Withdraw IP | 6 | 10 | 9
  TEAE with Fatal Outcome | 4 | 12 | 3
  Treatment Related TEAE with Fatal Outcome | 0 | 4 | 1

6. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment
Description: The discontinuation rate was defined as the percentage of participants who had study drug discontinued and was assessed throughout the conduct of the study.
Time Frame: Up to 30 Aug 2017 for CC-486 + nab-paclitaxel and 26 Nov 2019 for nab-paclitaxe and 20 Jul 2023 for Durva + nab-paclitaxel (up to 445 weeks)
Population: Safety Population included all participants who were randomized and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel
Number analyzed (Participants) | 79 | 78 | 79
percentage of participants | 100.0 | 100.0 | 100.0

7. Secondary Outcome: Dose Intensity Per Week of Nab-Paclitaxel
Description: Dose intensity was the cumulative dose divided by the dosing period in weeks.
Time Frame: as for outcome 2
Population: The treated population consisted of all participants who were randomized or assigned and received at least 1 dose of IP.
Measure: Mean (Standard Deviation); unit: mg/m^2/week
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel Alone
Number analyzed (Participants) | 79 | 78 | 79
mg/m^2/week | 54.73 (11.390) | 57.18 (13.605) | 58.61 (14.893)

8. Secondary Outcome: Dose Intensity Per Week of CC-486
Description: Dose intensity was the cumulative dose divided by the dosing period in weeks.
Time Frame: as for outcome 2
Population: The treated population consisted of all participants who randomized or assigned and received at least 1 dose of IP.
Measure: Mean (Standard Deviation); unit: mg/ week
Arm/Group | Nab-Paclitaxel + CC-486
Number analyzed (Participants) | 79
mg/ week | 716.66 (220.945)

9. Secondary Outcome: Dose Intensity Per Week of Durvalumab
Description: Dose intensity was the cumulative dose divided by the dosing period in weeks.
Time Frame: as for outcome 2
Population: The treated population consisted of all participants who randomized or assigned and received at least 1 dose of investigational Product.
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | Nab-Paclitaxel + Durvalumab
Number analyzed (Participants) | 77
mg/week | 279.96 (97.304)

10. Secondary Outcome: Percentage of Participants With Study Drug Dose Reductions
Description: A dose reduction occurred when the dose assigned at a visit was lower than the dose assigned at the previous visit. Dose reductions were typically caused by clinically significant laboratory abnormalities and/or treatment emergent adverse events or toxicities.
Time Frame: Up to 16 Jan 2017 for CC-486 + nab-paclitaxel and up to 26 Nov 2019 for nab-paclitaxel and Durva + nab-paclitaxel (up to 255 weeks)
Population: Safety Population included all participants who were randomized and received at least 1 dose of study drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel Alone
Number analyzed (Participants) | 79 | 78 | 79
Percentage of Participants
  Nab-Paclitaxel | 10.1 | 14.1 | 10.1
  CC-486: number analyzed (Participants) | 79 | 0 | 0
  CC-486 | 20.3 |  |
  Durvalumab (Reductions Not Allowed per Protocol): number analyzed (Participants) | 0 | 78 | 0
  Durvalumab (Reductions Not Allowed per Protocol) |  | 0.0 |

ADVERSE EVENTS:
Time Frame: SAEs and AEs were collected up to 4 weeks after receiving last dose of investigational product (IP) for nab-paclitaxel and CC-486 + nab-paclitaxel, and up to 90 days after the last IP dose for Durva + nab-paclitaxel; (Up to 354 weeks). Participants were assessed for all-cause mortality from their first dose to study completion (Up to 449 weeks).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Nab-Paclitaxel + CC-486 | Nab-Paclitaxel + Durvalumab | Nab-Paclitaxel
All-Cause Mortality (participants affected / at risk) | 62/81 | 48/79 | 50/80
Serious Adverse Events (participants affected / at risk) | 30/79 | 44/78 | 30/79
Other Adverse Events (participants affected / at risk) | 77/79 | 75/78 | 75/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel + CC-486 (N=79) | Nab-Paclitaxel + Durvalumab (N=78) | Nab-Paclitaxel (N=79)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 3 | 0
Retinal vasculitis (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Death (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 2 | 2 | 1
Performance status decreased (General disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 3 | 2 | 1
Sudden death (General disorders) | 1 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 3 | 1
Lung infection (Infections and infestations) | 0 | 2 | 0
Pelvic infection (Infections and infestations) | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 9 | 3
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 2 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel + CC-486 (N=79) | Nab-Paclitaxel + Durvalumab (N=78) | Nab-Paclitaxel (N=79)
Anaemia (Blood and lymphatic system disorders) | 12 | 27 | 24
Leukopenia (Blood and lymphatic system disorders) | 5 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 15 | 14 | 10
Vertigo (Ear and labyrinth disorders) | 4 | 2 | 3
Hypothyroidism (Endocrine disorders) | 0 | 6 | 0
Vision blurred (Eye disorders) | 4 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 3 | 8
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5 | 2
Constipation (Gastrointestinal disorders) | 32 | 21 | 26
Diarrhoea (Gastrointestinal disorders) | 33 | 30 | 20
Dyspepsia (Gastrointestinal disorders) | 5 | 5 | 6
Haemorrhoids (Gastrointestinal disorders) | 4 | 1 | 0
Nausea (Gastrointestinal disorders) | 45 | 19 | 20
Stomatitis (Gastrointestinal disorders) | 8 | 6 | 8
Vomiting (Gastrointestinal disorders) | 42 | 10 | 18
Asthenia (General disorders) | 26 | 36 | 25
Chills (General disorders) | 0 | 2 | 4
Fatigue (General disorders) | 24 | 22 | 23
General physical health deterioration (General disorders) | 4 | 4 | 1
Non-cardiac chest pain (General disorders) | 3 | 6 | 5
Oedema peripheral (General disorders) | 12 | 13 | 15
Pyrexia (General disorders) | 10 | 13 | 7
Bronchitis (Infections and infestations) | 2 | 2 | 4
Lower respiratory tract infection (Infections and infestations) | 1 | 12 | 3
Nasopharyngitis (Infections and infestations) | 5 | 4 | 5
Oral candidiasis (Infections and infestations) | 5 | 3 | 4
Respiratory tract infection (Infections and infestations) | 2 | 10 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 21 | 8
Urinary tract infection (Infections and infestations) | 2 | 10 | 4
Alanine aminotransferase increased (Investigations) | 2 | 4 | 0
Blood creatinine increased (Investigations) | 0 | 5 | 1
Neutrophil count decreased (Investigations) | 5 | 0 | 4
Weight decreased (Investigations) | 9 | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 27 | 27 | 24
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 5 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 5 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 10 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 10 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 8 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 5 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 4 | 8
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 9 | 4
Dizziness (Nervous system disorders) | 8 | 6 | 9
Headache (Nervous system disorders) | 9 | 10 | 10
Paraesthesia (Nervous system disorders) | 10 | 2 | 3
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 19 | 25 | 22
Anxiety (Psychiatric disorders) | 5 | 2 | 4
Depressed mood (Psychiatric disorders) | 0 | 4 | 1
Insomnia (Psychiatric disorders) | 9 | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 22 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 23 | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 11 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 26 | 21
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Flushing (Vascular disorders) | 1 | 0 | 4
Hypotension (Vascular disorders) | 2 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (7):
  • Study Protocol: ABI_007-NSCL_Protocol_AM5_Redacted_09December 2016 (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT02250326/Prot_001.pdf
  • Study Protocol: ABI-007-NSCL-006_Protocol_AM4_Redacted.31May2016 (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT02250326/Prot_002.pdf
  • Study Protocol: ABI_007-NSCL_Protocol_AM3_Redacted_14 April 2016 (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT02250326/Prot_003.pdf
  • Study Protocol: ABI_007-NSCL_Protocol_AM2_Redacted_18July2014 (2014-07-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT02250326/Prot_004.pdf
  • Study Protocol: ABI_007-NSCL_Protocol_AM1_Redacted_24 June 2014 (2014-06-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT02250326/Prot_005.pdf
  • Study Protocol: ABI_007-NSCL_Protocol_Original_Redacted_29May2014 (2014-05-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT02250326/Prot_006.pdf
  • Statistical Analysis Plan (2016-08-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT02250326/SAP_000.pdf